CLINICAL TRIAL: NCT04323592
Title: Prolonged Low Doses of Methylprednisolone for Patients With COVID-19 Severe Acute Respiratory Syndrome
Brief Title: Methylprednisolone for Patients With COVID-19 Severe Acute Respiratory Syndrome
Acronym: MP-C19
Status: Completed | Type: Observational
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, marco confalonieri, Head of Pulmonology and Critical care Dept., University of Trieste
Other Study IDs: MP-19 023_2020
Record Dates: First submitted 2020-03-19; First posted 2020-03-26 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Severe Acute Respiratory Syndrome (SARS) Pneumonia; Coronavirus Infections; ARDS, Human
Keywords: SARS-CoV-2,; SARS; ARDS; Methylprednisolone
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Pneumonia; Coronavirus Infections; Respiratory Distress Syndrome | interventions — Methylprednisolone; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: None Retained — Previous specific informed consent, blood samples of some patients treated with methylprednisolone were collected, in order to have the possibility to do
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed to Methylprednisolone: Consecutive SARS-CoV-2 positive patients with severe acute respiratory syndrome treated with methylprednisolone (MP) at low prolonged dose, fulfilling inclusion and exclusion criteria.
  Interventions: Drug: Methylprednisolone; Other: standard care
- Non-exposed to Methylprednisolone: Concurrent patients fulfilling the same inclusion and exclusion criteria, never treated with steroids.
  Interventions: Other: standard care

INTERVENTIONS:
Drug: Methylprednisolone — Usual standard of care plus Methylprednisolone (MP) 80 mg/kg IV bolus, followed by MP infusion of 80 mg/day in 240 mL normal saline at 10 mL/h. The infusion is continued for at least eight days and until achieving either a PaO2:FiO2 > 350 mmHg or a CRP < 20 mg/L. Treatment is then switched to oral administration of Methylprednisolone 16 mg or 20 mg IV twice daily until CRP returns to < 20% of normal range and/or PaO2:FiO2 > 400 or SatHbO2 ≥ 95%. The decision to apply the protocol to Covid-19 is left to the discretion of the treating team for each individual patient.
  Groups: Exposed to Methylprednisolone
Other: standard care — usual standard of care:
  * oxygen therapy (regular or high-flow) and monitoring
  * empiric antibiotic therapy
  * mechanical ventilation (invasive or noninvasive)
  * ECMO when needed and available
  * pronation when possible
  * other treatment which can be used are: antivirals, chloroquine, vitamins

SUMMARY:
COVID-19 infection is overwhelming Italian healthcare. There is an urgent need for a solution to the lack of ICU beds and increasing deaths day after day.

A recent retrospective Chinese paper (JAMA Intern Med, online March 13, 2020) showed impressive positive effect of methylprednisolone (MP) on survival of SARS-CoV-2 critically ill patients. Moreover, the Italian Infectious Disease leading institution guidelines for COVID-19 clinical management included as an option for patients with "incipient worsening of respiratory functions" methylprednisolone treatment at an approximate dose of 80mg.

The main objective of this multi-centre observational trial is to analyse the association of low dose prolonged infusion of methylprednisolone (MP) for patients with severe acute respiratory syndrome with composite primary end-point (ICU referral, need for intubation, in-hospital death at day 28).

DETAILED DESCRIPTION:
Comparison of two groups of patients SARS-CoV-2 positive with severe acute respiratory syndrome:

1. Exposed to low prolonged doses of Methylprednisolone
2. Not exposed to corticosteroids (standard of care alone)

The two group will be weighted by means of a propensity score according to:

1. Sex
2. Age
3. C-reactive protein (CRP) at baseline
4. Sequential Organ Failure Assessment (SOFA) score at baseline
5. PaO2/FiO2 ratio at baseline (ratio of arterial oxygen partial pressure to fractional inspired oxygen)

Anti-viral agents, chloroquine, respiratory support (any), and antibiotics (any) are allowed in each study group. Corticosteroids use, other than per-protocol Methylprednisolone in the exposed group is a reason for dropout.

1. The exposed group is treated with Methylprednisolone at study entry (baseline) according to a protocol based on the Italian national recommendations for COVID-19 management: a loading dose of 80 mg IV, followed by an infusion of 80 mg/day in 240 mL normal saline at 10 mL/h. The infusion is continued for at least eight days and until achieving either a PaO2:FiO2 > 350 mmHg or a CRP < 20 mg/L. Treatment is then switched to oral administration of Methylprednisolone 16 mg or 20 mg IV twice daily until CRP returns to < 20% of normal range and/or PaO2:FiO2 > 400 or SatHbO2 ≥ 95%. The decision to apply the protocol to Covid-19 is left to the discretion of the treating team for each individual patient.
2. Unexposed patients will be selected from concurrent consecutive COVID-19 patients with the same inclusion and exclusion criteria and blinded to outcome data.

ELIGIBILITY:
Inclusion Criteria:

1. SARS-CoV-2 positive
2. Age >17 years and < 80 years
3. P/F < 250 mmHg
4. Bilateral pneumonia (infiltrates/interstitial)
5. CRP >10mg/dL (or >100mg/L)
6. Alternatively to 4-5-6 criteria a diagnosis of ARDS according to the Berlin definition (Ranieri M, et al. JAMA 2012)

Exclusion Criteria:

* Heart failure as predominant cause of acute respiratory failure
* Decompensated liver cirrhosis
* Cancer
* Organ transplantation
* HIV+
* dialysis
* long-term oxygen therapy, home mechanical ventilation
* Idiopathic pulmonary fibrosis
* Progressive neuromuscular disorders (e.g. Duchenne, Pompe, ALS)
* Dementia or decompensated psychiatric diseases
* immunosuppressive treatments
* Chronic use of corticosteroids
* Use of Tocilizumab
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to Respiratory High dependency units for severe acute respiratory syndrome associated to COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Confalonieri, MD, Principal Investigator — University of Trieste
Locations (1):
- Marco Confalonieri, Trieste, TS, Italy

IPD SHARING:
Plan to Share IPD: No
Anonymised data will be available only to data manager who can visualise clinical chart anytime when is needed

REFERENCES:
- [Background] Nicastri E, Petrosillo N, Ascoli Bartoli T, Lepore L, Mondi A, Palmieri F, D'Offizi G, Marchioni L, Murachelli S, Ippolito G, Antinori A. National Institute for the Infectious Diseases "L. Spallanzani", IRCCS. Recommendations for COVID-19 clinical management. Infect Dis Rep. 2020 Mar 16;12(1):8543. doi: 10.4081/idr.2020.8543. eCollection 2020 Feb 25. PMID 32218915
- [Derived] Salton F, Confalonieri P, Meduri GU, Santus P, Harari S, Scala R, Lanini S, Vertui V, Oggionni T, Caminati A, Patruno V, Tamburrini M, Scartabellati A, Parati M, Villani M, Radovanovic D, Tomassetti S, Ravaglia C, Poletti V, Vianello A, Gaccione AT, Guidelli L, Raccanelli R, Lucernoni P, Lacedonia D, Foschino Barbaro MP, Centanni S, Mondoni M, Davi M, Fantin A, Cao X, Torelli L, Zucchetto A, Montico M, Casarin A, Romagnoli M, Gasparini S, Bonifazi M, D'Agaro P, Marcello A, Licastro D, Ruaro B, Volpe MC, Umberger R, Confalonieri M. Prolonged Low-Dose Methylprednisolone in Patients With Severe COVID-19 Pneumonia. Open Forum Infect Dis. 2020 Sep 12;7(10):ofaa421. doi: 10.1093/ofid/ofaa421. eCollection 2020 Oct. PMID 33072814

RESULTS

PARTICIPANT FLOW:
Groups:
- Exposed to Methylprednisolone: SARS-CoV-2 positive patients with severe acute respiratory syndrome consecutively treated with methylprednisolone (MP) at prolonged dose.
  Inclusion criteria checked, the patient undergo 80mg iv bolus of MP followed by infusion (10cc/h) of MP in 240cc 0.9% saline every day until PaO2/FiO2 increase over 350 and/or CRP decrease below 20mg/L, then MP is administered PO tapering slowly until normal CRP values (+20%) are reached.
  Methylprednisolone: after initial 80mg iv bolus followed by 80mg in 240cc 0.9% saline administered iv at 10cc/h speed for at least 7 day or more. Duration of Methylprednisolone treatment depends from CRP and P/F values already described in arm/group description
  standard care: usual standard of care:
  * respiratory support
  * empiric antibiotic therapy
  * mechanical ventilation (invasive or noninvasive)
  * pronation when possible
  * other treatment which can be used are: antivirals, chloroquine, vitamins
- Non-exposed to Methylprednisolone: Concurrent patients with the same inclusion/section exclusion criteria never treated with steroids, strictly matched according to gender and age (+/-10 years) and other three parameters:
  CRP, SOFA score, PaO2:FiO2 -> each parameter must be <20% difference between case and control.
  standard care: usual standard of care:
  * respiratory support
  * empiric antibiotic therapy
  * mechanical ventilation (invasive or noninvasive)pronation when possible
  * other treatment which can be used are: antivirals, chloroquine, vitamins
Period: Overall Study
Arm/Group | Exposed to Methylprednisolone | Non-exposed to Methylprednisolone
Started | 83 | 90
Completed | 83 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exposed to Methylprednisolone: SARS-CoV-2 positive patients with severe acute respiratory syndrome consecutively treated with methylprednisolone (MP) at low prolonged dose.
  At admission, inclusion criteria checked, the patient undergo 80mg iv bolus of MP followed by infusion (10cc/h) of MP in 240cc 0.9% saline every day until PaO2/FiO2 increase over 350 and/or CRP decrease below 20mg/L, then MP is administered PO tapering until normal CRP values (+20%) are reached.
  Methylprednisolone: Methylprednisolone given at low prolonged dose infusion after initial 80mg iv bolus at admission followed by 80mg in 240cc 0.9% saline administered iv at 10cc/h speed for at least 7 day or more. Duration of Methylprednisolone treatment depends from CRP and P/F values already described in arm/group description
  standard care: usual standard of care:
  * oxygen therapy (regular or high-flow) and monitoring
  * empiric antibiotic therapy
  * mechanical ventilation (invasive or noninvasive)
  * ECMO when needed and available
  * pronati
- Non-exposed to Methylprednisolone: Concurrent patients with the same inclusion/section exclusion criteria never treated with steroids, strictly matched according to gender and age (+/-10 years) and other three parameters:
  CRP, SOFA score, PaO2:FiO2 -> each parameter must be <20% difference between case and control.
  standard care: usual standard of care:
  * oxygen therapy (regular or high-flow) and monitoring
  * empiric antibiotic therapy
  * mechanical ventilation (invasive or noninvasive)
  * ECMO when needed and available
  * pronation when possible
  * other treatment which can be used are: antivirals, chloroquine, vitamins
- Total: Total of all reporting groups
Arm/Group | Exposed to Methylprednisolone | Non-exposed to Methylprednisolone | Total
Number analyzed (Participants) | 83 | 90 | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 34 | 69
  >=65 years | 48 | 56 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.39 (10.73) | 67.08 (8.24) | 65.79 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 53
  Male | 54 | 66 | 120
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 83 | 90 | 173
C-reactive Protein [Mean (Standard Deviation); unit: mg/L] | 136.92 (72.57) | 148.64 (75.59) | 143.01 (74.17)
PaO2/FiO2 [Mean (Standard Deviation); unit: ratio] | 152.02 (49.84) | 151.01 (60.26) | 151.50 (55.35)
Sequential Organ Failure Assessment (SOFA) Score [Median (Inter-Quartile Range); unit: score] — Sum of subscales scoring the function of: nervous system, kidneys, coagulation, respiratory system, cardiovascular system, liver.
  Values ranging 0-24; higher values represent worse outcome.
  score | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
Lactates [Mean (Standard Deviation); unit: mmol/L] | 1.76 (1.97) | 1.34 (0.51) | 1.52 (1.32)
Lymphocytes [Mean (Standard Deviation); unit: cells/uL] | 622.28 (650.62) | 954.5 (914.7) | 938.94 (797.81)
D-dimer [Median (Inter-Quartile Range); unit: ug/L Fibrinogen Equivalent Units (FEU)] | 780 [530 to 1207] | 890 [506.75 to 1757] | 813 [518 to 1560.5]
lactate dehydrogenase (LDH) [Mean (Standard Deviation); unit: U/L] | 380 (132.93) | 413.06 (143.83) | 396.41 (138.96)
Respiratory rate [Mean (Standard Deviation); unit: Breaths per minute] | 23.74 (5.95) | 25.27 (6.76) | 24.55 (6.41)

OUTCOME MEASURES:

1. Primary Outcome: Composite Primary End-point: Admission to ICU, Need for Invasive Mechanical Ventilation (MV), or All-cause Death by Day 28
Description: We reported below the number of participants meeting at least one of three among death or ICU admission or Invasive mechanical ventilation.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed to Methylprednisolone | Non-exposed to Methylprednisolone
Number analyzed (Participants) | 83 | 90
Participants | 19 | 40

2. Primary Outcome: In-hospital Death Within 28 Days
Description: We reported below the number of participants who died within 28 days, during the hospital stay.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed to Methylprednisolone | Non-exposed to Methylprednisolone
Number analyzed (Participants) | 83 | 90
Participants | 6 | 21

3. Primary Outcome: Admission to Intensive Care Unit (ICU)
Description: We reported below the number of participants admitted to ICU within 28 days.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed to Methylprednisolone | Non-exposed to Methylprednisolone
Number analyzed (Participants) | 83 | 90
Participants | 15 | 27

4. Primary Outcome: Endotracheal Intubation (Invasive Mechanical Ventilation)
Description: We reported below the number of participants who needed endotracheal intubation during ICU admission
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed to Methylprednisolone | Non-exposed to Methylprednisolone
Number analyzed (Participants) | 83 | 90
Participants | 15 | 26

5. Secondary Outcome: Change in C-reactive Protein (CRP)
Description: Change in C-reactive protein after 7 days from baseline. A reduction of CRP reveals a laboratory improvement.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Exposed to Methylprednisolone | Non-exposed to Methylprednisolone
Number analyzed (Participants) | 83 | 90
mg/L | -82.08 (28.24) | -34.34 (66.64)

6. Secondary Outcome: Number of Days Free From Mechanical Ventilation
Description: number of days free from mechanical ventilation (both invasive and non-invasive) by day 28
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Exposed to Methylprednisolone | Non-exposed to Methylprednisolone
Number analyzed (Participants) | 83 | 90
days | 19.11 (8.73) | 14.34 (11.65)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Exposed to Methylprednisolone | Non-exposed to Methylprednisolone
All-Cause Mortality (participants affected / at risk) | 9/83 | 24/90
Serious Adverse Events (participants affected / at risk) | 6/83 | 9/90
Other Adverse Events (participants affected / at risk) | 23/83 | 21/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exposed to Methylprednisolone (N=83) | Non-exposed to Methylprednisolone (N=90)
Shock (General disorders) | 0 (0) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 2 (2) | 4 (4)
Disseminated intravascular coagulation (Vascular disorders) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exposed to Methylprednisolone (N=83) | Non-exposed to Methylprednisolone (N=90)
Bacterial superinfection (General disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 9 (9) | 2 (2)
Hyperglycemia (Endocrine disorders) | 8 (8) | 0 (0)
Hypokalemia (General disorders) | 6 (6) | 13 (13)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Transaminase elevation (Hepatobiliary disorders) | 2 (2) | 2 (2)
QT elongation (Cardiac disorders) | 7 (7) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Informed Consent Form (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT04323592/ICF_003.pdf
  • Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT04323592/SAP_004.pdf
  • Study Protocol (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT04323592/Prot_006.pdf